CLINICAL TRIAL: NCT07009782
Title: Evaluation of the Postoperative Analgesic Efficacy of the Quadroiliac Plane (QIP) Block in Femur Fracture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, anesthesiology and reanimation specialist, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QIPB in femur fractures
Record Dates: First submitted 2025-05-28; First posted 2025-06-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Femur Fracture
Keywords: Postoperative Pain
MeSH Terms: conditions — Femoral Fractures; Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Pain assessments, including Numerical Rating Scale (NRS) scores, cold test evaluations, and Quality of Recovery-15 (QOR-15) questionnaires, will be performed by outcome assessors who are blinded to the group allocation. These assessors will not be involved in the administration of the Quadroiliac Plane (QIP) block and will be unaware of whether the patient received the block or not. This ensures unbiased evaluation of analgesic outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QIP Block Group (Experimental): Participants in this group will receive a Quadroiliac Plane (QIP) block using 40 mL of 0.25% bupivacaine under ultrasound guidance, applied postoperatively while in the prone position. The block will be performed only on the surgical side. All patients will also receive standard postoperative multimodal analgesia, including intravenous patient-controlled analgesia (PCA) with fentanyl.
  Interventions: Procedure: QIP block
- Control Group (No Intervention): Participants in this group will not receive a regional block. They will be managed with standard postoperative multimodal analgesia, including intravenous patient-controlled analgesia (PCA) with fentanyl.

INTERVENTIONS:
Procedure: QIP block — The Quadroiliac Plane (QIP) block is a novel ultrasound-guided fascial plane block. In this study, it will be performed postoperatively under spinal anesthesia in the prone position. A low-frequency convex transducer will be used to visualize the quadratus lumborum muscle at its attachment to the inner iliac crest. Using an in-plane technique with a 22G x 100 mm needle, 40 mL of 0.25% bupivacaine will be injected into the fascial plane beneath the quadratus lumborum muscle. The block will be performed unilaterally on the surgical side. The aim is to provide postoperative analgesia in patients undergoing femur fracture surgery.
  Arms: QIP Block Group

SUMMARY:
The goal of this clinical trial is to learn whether the Quadroiliac Plane (QIP) block helps reduce postoperative opioid use in adults undergoing femur fracture surgery. It will also evaluate the pain control effectiveness, dermatomal spread, and safety of the QIP block. The main questions it aims to answer are:

Does the QIP block reduce total opioid (fentanyl) consumption within 24 hours after surgery?

Does the QIP block reduce the need for rescue analgesia?

What is the extent of dermatomal spread and are there any side effects or complications?

Researchers will compare patients receiving the QIP block to those receiving standard care without a block to see if the QIP block improves pain management outcomes.

Participants will:

Undergo femur fracture surgery under spinal anesthesia

Be randomly assigned to receive either the QIP block or no block after surgery

Use a patient-controlled analgesia (PCA) device with fentanyl

Have their pain scores, drug use, and recovery quality measured over 24 hours

Undergo a cold test at 2 hours post-op and complete a recovery questionnaire at 24 hours

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, single-center clinical trial designed to evaluate the postoperative analgesic efficacy of the Quadroiliac Plane (QIP) block in patients undergoing femur fracture surgery, specifically partial hip arthroplasty under spinal anesthesia. The primary objective of the study is to assess the impact of the QIP block on total opioid consumption (fentanyl via PCA) during the first 24 hours postoperatively. Secondary objectives include evaluation of rescue analgesia needs, dermatomal spread of the block, incidence of motor block or complications, block feasibility and application time, patient satisfaction, and length of hospital stay.

Eligible participants aged 18 years or older who are scheduled for elective partial hip arthroplasty due to femoral neck fracture and meet inclusion criteria will be invited to participate. After obtaining written informed consent, patients will be randomly assigned to one of two groups using a computer-generated sequence and sealed envelope method. The intervention group will receive a QIP block postoperatively using 40 mL of 0.25% bupivacaine under ultrasound guidance. The control group will receive no regional block. Both groups will receive standard postoperative multimodal analgesia, including intravenous patient-controlled analgesia (PCA) with fentanyl.

Pain will be assessed using the Numerical Rating Scale (NRS), which ranges from 0 (no pain) to 10 (worst imaginable pain), at rest and with movement at 0, 6, 12, and 24 hours postoperatively. Rescue analgesia (50 mg dexketoprofen IV over 20 minutes) will be administered if needed. The dermatomal spread of the block will be evaluated using an alcohol-based cold test at 2 hours postoperatively. At 24 hours, all patients will complete the Quality of Recovery-15 (QOR-15) questionnaire, which scores recovery from 0 (poor recovery) to 150 (excellent recovery).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Scheduled for partial hip arthroplasty due to femur fracture
* ASA physical status classification I to III
* No contraindications to regional anesthesia or study medications
* Capable of understanding and using patient-controlled analgesia (PCA)
* Provided written informed consent

Exclusion Criteria:

* ASA classification IV or higher
* History of bleeding disorders or use of anticoagulant therapy
* Known allergy to local anesthetics
* Presence of neuropathic pain disorders
* Undergoing emergency surgery
* Unable to operate PCA device
* Declined to participate or refused consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Total Opioid Consumption Within the First 24 Hours Postoperatively | 24 hours postoperatively
  The total amount of fentanyl (in micrograms) administered via intravenous patient-controlled analgesia (PCA) will be recorded during the first 24 hours after surgery. This will be used to assess the analgesic efficacy of the Quadroiliac Plane (QIP) block compared to standard care without a block.

SECONDARY OUTCOMES:
Rescue Analgesia Requirement | 24 hours
  The number of patients who require additional rescue analgesia (50 mg intravenous dexketoprofen) within the first 24 hours postoperatively will be recorded.
Pain Scores at Rest and on Movement | 0,6,12 and 24 hours
  Pain intensity will be measured using the Numerical Rating Scale (NRS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Assessments will be conducted both at rest and during movement at 0, 6, 12, and 24 hours after surgery. Higher scores indicate worse pain.
Extent of Dermatomal Coverage Measured by Cold Sensation Response to Alcohol Swab at 2 Hours Post-QIP Block | 2 hours postoperatively
  Dermatomal spread will be assessed using an alcohol-based cold test 2 hours after administration of the Quadroiliac Plane (QIP) Block. A trained clinician will apply alcohol-soaked gauze to the skin in a cranio-caudal direction along the abdomen and hip region. The patient will be asked to report changes in cold sensation compared to unblocked areas. The lowest and highest dermatomes with altered cold sensation (reduced or absent) will be recorded for each side.
Postoperative Recovery Quality | 24 hours postoperatively
  Patients will complete the Quality of Recovery-15 (QoR-15) questionnaire 24 hours after surgery to evaluate their postoperative recovery experience. The QoR-15 consists of 15 items, each scored from 0 to 10, resulting in a total score range of 0 to 150. Higher scores indicate better recovery and a more favorable patient-reported outcome
Block-Related Complications | 24 hours
  Any complications or side effects related to the QIP block (e.g., motor block, hematoma, infection) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Engin ihsan Turan, Specialist, Principal Investigator — Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Turan EI, Baydemir AE, Sahin AS. Efficacy of the quadro-iliac plane block in postoperative pain management for proximal femoral nail surgeries. Minerva Anestesiol. 2025 Mar;91(3):221-223. doi: 10.23736/S0375-9393.24.18506-9. Epub 2024 Nov 4. No abstract available. PMID 39495169